CLINICAL TRIAL: NCT05456724
Title: A 3-Part, First-in-human, Double-Blind, Randomized, and Placebo-Controlled Study Assessing the Safety, Tolerability, and Efficacy of TO-O-1001 Ophthalmic Solution in Healthy Subjects and in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: A Study to Investigate the Effect of IOP-lowering With TO-O-1001 Eye Drops in Healthy Subjects and in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theratocular Biotek Co. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Organization: Metagone Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TO-01C101
Record Dates: First submitted 2022-06-27; First posted 2022-07-13 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (TO-O-1001) (Experimental): Drug: TO-O-1001 Dose level: 0.05% and 0.1% Dosage form: ophthalmic solution Route of administration: topical ocular
  Interventions: Drug: TO-O-1001
- B (Placebo) (Placebo Comparator): Dosage form: ophthalmic solution Route of administration: topical ocular
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TO-O-1001 — TO-O-1001 ophthalmic solution in two concentration (0.05% and 0.1%) ocular administration only one drop in one eye
  Arms: A (TO-O-1001)
Other: Placebo — The placebo is of same visual appearance and identical formulation as TO-O-1001, except the active component TO-168 ocular administration only one drop in one eye
  Arms: B (Placebo)

SUMMARY:
This is a Phase I/II stage to investigate the safety, tolerability, and ocular hypotensive efficacy of TO-O-1001 in healthy volunteers and patients with Open-Angle Glaucoma or Ocular Hypertension.

The proposed trial consists of 3 study parts to be conducted at Nucleus Network Melbourne.

This study will enroll up to 34 evaluable healthy volunteers in part 1(SAD) and part 2(MD) and 16 evaluable patients with Open-Angle Glaucoma or Ocular Hypertension in part 3(MD).

Note- As of 14Mar2023, enrolment has been completed for Part 1 and Part 2 and recruitment is pending now for Part 3.

ELIGIBILITY:
Inclusion Criteria:

For Healthy Subjects (Parts 1 & 2)

1. 18 - 59-year-old healthy male or female subjects who are non-lactating and non-pregnant.
2. BMI 18.0~32.0(kg/m2) and body weight more than 45kg.
3. Intraocular pressure between 10 - 21 mm Hg (inclusive) in each eye.
4. Best-corrected visual acuity (BCVA) in each eye of 20/40 ETRDS or better.
5. The informed consent form has been read, signed and dated by the subjects.
6. Able to communicate well with the investigator and comply with the requirements of the study.

For Patients (Part 3)

1. Must be 18 years of age or older.
2. Diagnosis of primary open angle glaucoma (POAG) or ocular hypertension (OHT).
3. Unmedicated or after washout intraocular pressure (IOP) >20 mmHg and < 30 mmHg in study eye at T0 (T0 = 08:00AM~10:00 AM) of the first qualification visit (Day 1).
4. Best-corrected visual acuity (BCVA) equivalent to 20/200 ETRDS or better.
5. The informed consent form has been read, signed and dated by the subjects.
6. Able to communicate well with the investigator and comply with the requirements of the study

Exclusion Criteria:

For Healthy Subjects (Parts 1 & 2)

1. Subjects has chronic or acute ophthalmic disease including glaucoma, macular degeneration, and clinically significant cataract (primary or secondary).
2. Subjects has previous glaucoma intraocular surgery or glaucoma laser procedures within 3 years.
3. Subjects has refractive surgery (e.g., radial keratotomy, PRK, LASIK, etc.) within 5 years.
4. Subjects has ocular trauma within the past 6 months, or ocular surgery or laser treatment within the past three months (e.g., laser treatment for glaucoma or retina).

For Patients (Part 3)

1. Closed or very narrow angles (Grade 0-1) or those the investigator judges as occludable and/or with evidence of peripheral anterior synechiae (PAS) ≥ 180 degrees by gonioscopy within 6 months prior to Screening Visit in either eye. (Patent laser iridotomy with Grade 1-2 angles is acceptable in either eye, providing the PAS criteria are still met).
2. Previous glaucoma intraocular surgery in either eye. Prior laser trabeculoplasty (ALT or SLT) in either eye is allowed if performed more than 6 months prior to Screening Visit.
3. Any non-glaucoma intraocular surgery within 3 months prior to Screening Visit in either eye.
4. Participation in a clinical study with use of any investigational drug or treatment within 28 days prior to Baseline (Day 1).
5. Clinically significant abnormalities in: laboratory tests, physical examination, vital signs and/or ECG at Screening Visit. If in the investigator's judgment a subjects with clinically significant abnormalities is appropriate for enrollment in the study, a discussion between the investigator and the Medical Monitor must occur and be documented prior to enrollment of this subjects in the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of TO-O-1001 though the incidence of adverse events. | Up to 28 days
  Number of participants with treatment-emergent adverse events (AEs).
Evaluate the ocular hypotensive efficacy of TO-O-1001 through Goldmann Applanation Tonometry. | Up to 28 days
  The primary efficacy outcome is mean IOP.

SECONDARY OUTCOMES:
Pharmacokinetics of TO-O-1001. Blood samples obtained to evaluate the systemic exposure. | Up to 8 days
  Parameter: Area Under the Curve (AUC)
Pharmacokinetics of TO-O-1001. Blood samples obtained to evaluate the systemic exposure. | Up to 8 days
  Parameter: Maximum Concentration
Pharmacokinetics of TO-O-1001. Blood samples obtained to evaluate the systemic exposure. | Up to 8 days
  Parameter: Maximum observed concentration (Cmax in first and last dose)
Pharmacokinetics of TO-O-1001. Blood samples obtained to evaluate the systemic exposure. | Up to 8 days
  Parameter: Area under the concentration-time curve (AUC0-t and AUC0-inf in first and last dose)
Pharmacokinetics of TO-O-1001. Blood samples obtained to evaluate the systemic exposure. | Up to 8 days
  Parameter: Time of observed Cmax
Pharmacokinetics of TO-O-1001. Blood samples obtained to evaluate the systemic exposure. | Up to 8 days
  Parameter: Terminal elimination half-life and elimination constant in first and last dose
Best Corrected Visual Acuity (BCVA) of TO-O-1001. | Up to 28 days
  Visual function of the study eye was assessed using the ETDRS protocol. A higher score represents better functioning.
Safety and tolerability of TO-O-1001 through the incidence, severity and causality of serious adverse events (SAEs). | Up to 28 days
  Number of participants with treatment-emergent serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Francis, Principal Investigator — Nucleus Network Melbourne
Locations (1):
- Nucleus Network Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No